CLINICAL TRIAL: NCT04403243
Title: COLchicine Versus Ruxolitinib and Secukinumab in Open-label Prospective Randomized Trial in Patients With COVID-19
Acronym: COLORIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lomonosov Moscow State University Medical Research and Educational Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSU080520
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: COVID 19
Keywords: COVID 19; colchicine; ruxolitinib; secukinumab
MeSH Terms: conditions — COVID-19 | interventions — Colchicine; ruxolitinib; secukinumab; Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 3:1:1:3 into four groups: colchicine, ruxolitinib, secukinumab, and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. Colchicine (Experimental): 30 Patients with mild and severe COVID 19 Patients will get investigated therapy for ten days. Patients will be follow-up during 45 days after randomization
  Interventions: Drug: Colchicine
- 2. Ruxolitinib (Experimental): 10 Patients with mild and severe COVID 19 Patients will get investigated therapy for ten days. Patients will be follow-up during 45 days after randomization
  Interventions: Drug: Ruxolitinib 5 MG
- 3.Secukinumab (Experimental): 10 Patients with mild and severe COVID 19 Patients will get investigated therapy singly. Patients will be follow-up during 45 days after randomization
  Interventions: Drug: Secukinumab 150 MG/ML Subcutaneous Solution [COSENTYX]
- 4.Standard treatment (Active Comparator): -30 patients Patients with mild and severe COVID 19 Patients will get investigated therapy for ten days. Patients will be follow-up during 45 days after randomization
  Interventions: Other: standard therapy

INTERVENTIONS:
Drug: Colchicine — 0.5mg twice a day per os during the first three days and then 0.5mg daily per os if weight < 86 kg or 0.5mg twice a day per os if weight > 85kg for seven days.
  Arms: 1. Colchicine
Drug: Ruxolitinib 5 MG — Ruxolitinib - 5mg twice a day per os for ten days
  Arms: 2. Ruxolitinib
Drug: Secukinumab 150 MG/ML Subcutaneous Solution [COSENTYX] — Secukinumab - 300mg subcutaneously singly
  Arms: 3.Secukinumab
Other: standard therapy — standard therapy for COVID 19
  Arms: 4.Standard treatment

SUMMARY:
Patients with mild and severe coronavirus disease 2019 (COVID 19) will be randomized 3:1:1:3 into four groups: colchicine, ruxolitinib, secukinumab, and control groups. . Patients will be follow-up during 45 days after randomization. Change in clinical assessment score COVID 19 (CAS COVID 19) between baseline and 12th day will be evaluated as the primary endpoint. Risk of death or mechanical ventilation during 45 days after randomization will also be assessed

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent
* COVID 19 with the mild and severe course. The diagnosis could be made with positive polymerase chain reaction (PCR) (International Statistical Classification (ICD-10) code - U07.1) and/or virus pneumonia in computer tomography (ICD 10 code - U07.2)
* Lung exposure on CT more than 25%
* Sp02 without supportive oxygen ≤ 93%
* C-reactive protein > 60 mg/l or elevation of C reactive protein 3 times in 8-14 days after first symptoms

Exclusion Criteria:

* pregnancy and breastfeeding
* hypersensitivity to colchicine
* hypersensitivity to ruxolitinib
* hypersensitivity to secukinumab
* Known liver failure
* Glomerular filtration rate <20 ml/ min
* physician judgment that the patient will need mechanical ventilation in 24 hours
* QTc > 450 ms
* other indications for to colchicine, ruxolitinib, and secukinumab
* Chronic therapy with corticosteroids or immunosuppressive therapy
* Active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-08-23 (Actual)

PRIMARY OUTCOMES:
change from baseline in clinical assessment score COVID 19 (CAS COVID 19) Frame: baseline | baseline, day 12
  CAS COVID 19 measures clinical and laboratory parameters in 7 domains:
  1. respiratory rate (< 18 - 0 point; 18-22 - 1 point; 23-26 - 2 point; >26 - 3 point)
  2. body temperature (35.5 - 37.0 - 0 point; < 35.5 - 1 point; 37.1 - 38.5 - 1 point; > 38.5 - 2 point)
  3. Sp02 without support oxygen (> 93% - 0 point; 90-93% - 1 point; < 90% - 2 point)
  4. ventilation (not required - 0 point; low-flow ventilation - 1 point; Non-invasive positive pressure ventilation - 2 point; mechanical ventilation - 3 point)
  5. C-reactive protein (> 10 - 0 point; 10-59 - 1 point; 60-120 - 2 point; > 120 - 3 point)
  6. d - dimer (< 0.51 - 0 point; 0.51 - 2.0 - 1 point; 2.01 - 5.0 - 2, > 5.0 - 3 point)
  7. exposure area on lung CT (no pneumonia - 0; 1-24% - 1 point; 25-50% - 2; 51-75% - 3, > 75% - 4).
  Minimal number of points - 0; max - 20. Lower the score-better health

SECONDARY OUTCOMES:
Combine endpoint: Time to death or mechanical ventilation | 45 days
  time to death or mechanical ventilation
C-reactive protein | baseline, day 12, day 45
  Change from baseline in C-reactive protein
D-dimer | baseline, day 12, day 45
  Change from baseline in D-dimer
EuroQol Group. EQ-5D™ | baseline, day 12, day 45
  Change from baseline in EQ-5D-3L™ The EQ-5D-3L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D-3L descriptive system comprises the 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box to the most appropriate statement. This decision results into a 1-digit number, . The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome by patient's own judgement.
exposure area on lung CT | baseline, day 12, day 45
  Change from baseline in exposure area on lung CT

CONTACTS AND LOCATIONS:
Locations (1):
- Lomonosov Moscow State University Medical Research and Educational Center, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 4 month
Access Criteria: Medical professionals By the request

REFERENCES:
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014